CLINICAL TRIAL: NCT05217927
Title: A Phase 4 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rimegepant in Episodic Migraine Prevention With Multiple Dosing Regimens
Brief Title: Efficacy and Safety Study of Rimegepant in Episodic Migraine Prevention With Multiple Dosing Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-404; 2021-005239-22 (EudraCT Number); C4951010 (Other: Alias Study Number)
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: Migraine; Episodic Migraine; Adult Migraine; Calcitonin Gene-related Peptide; Migraine Prevention; Migraine Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rimegepant 75mg Orally Disitegrating Tablet (ODT)daily dosing (Experimental): Double-blind Treatment Phase: Rimegepant 75 mg ODT dosed daily
  Open-Label Extension Phase:
  Rimegepant 75 mg ODT dosed daily
  Interventions: Drug: Rimegepant 75mg daily dosing
- Rimegepant 75mg Orally Disintegrating Tablet (ODT)every other day dosing (Experimental): Double-blind Treatment Phase: Rimegepant 75 mg ODT every other day dosing alternating with matching placebo
  Interventions: Drug: Rimegepant 75mg every other day dosing
- Placebo comparator dosing (Placebo Comparator): Double-blind Treatment Phase: matching placebo dosed daily
  Interventions: Drug: Placebo comparator dosing

INTERVENTIONS:
Drug: Rimegepant 75mg daily dosing — Daily
  Arms: Rimegepant 75mg Orally Disitegrating Tablet (ODT)daily dosing
Drug: Rimegepant 75mg every other day dosing — Every other day
  Arms: Rimegepant 75mg Orally Disintegrating Tablet (ODT)every other day dosing
Drug: Placebo comparator dosing — Placebo comparator
  Arms: Placebo comparator dosing

SUMMARY:
The purpose of this study is to compare the efficacy and safety of daily and every other day dosing of rimegepant to placebo as a preventive treatment for episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

1) Target Population: Subject has at least 1 year history of episodic migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:

1. Age of onset of migraines prior to 50 years of age
2. Migraine attacks, on average, lasting 4-72 hours if untreated
3. Per subject report, 4-14 migraine attacks per month within the last 3 months prior to the Screening Visit (month is defined as 4 weeks for the purpose of this protocol

Exclusion Criteria:

1. Sex and Reproductive Status:

   1. WOCBP who are unwilling or unable to use an acceptable contraceptive method or abstinence to avoid pregnancy for the entire study and for 60 days after the last dose of study drug
   2. Women who are pregnant or breastfeeding
   3. Women with a positive pregnancy test at screening or prior to study drug administration
2. Prohibited Medications:

   1. Use of prophylactic migraine medication within 30 days prior to the Screening Visit.
   2. History of use of analgesics (e.g., non-steroidal anti-inflammatory drugs [NSAIDs] or acetaminophen) on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit.
   3. Use of medication accepted for treatment of acute migraine for a nonmigraine indication on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit.
   4. Subjects who previously discontinued biologic migraine medication must have done so at least 6 months (24 weeks) prior to the Screening Visit.
   5. Subjects taking a prohibited medication as defined per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (107):
- United States (30):
  - AMR Clinical, Tempe, Arizona
  - Axiom Research, Llc, Colton, California
  - Clinical Research Institute, Los Angeles, California
  - Wr-Pri, Llc, Newport Beach, California
  - California Neuroscience Research Medical Group, inc., Sherman Oaks, California
  - Neurology Offices of South Florida, PLLC, Boca Raton, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Collective Medical Research, Overland Park, Kansas
  - Clinvest Research, LLC, Springfield, Missouri
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - Montefiore Medical Center, The Bronx, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Wellnow Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Huber Heights, Ohio
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research - Columbia, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Tribe Clinical Research LLC, Greenville, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - APD Clinical Research, Magnolia, Texas
  - Wasatch Clinical Research , LLC(Administrative Location), Salt Lake City, Utah
  - Seattle Clinical Research Center, Seattle, Washington
- Austria (2):
  - Medizinische Universitat Innsbruck, Innsbruck, Tyrol
  - Christian-Doppler-Klinik, Salzburg
- Canada (12):
  - Calgary Headache & Assessment Management Program (CHAMP), Calgary, Alberta
  - OCT Research ULC, Kelowna, British Columbia
  - James K. Lai MD Inc., Vancouver, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Manna Research Inc. (Burlington North), Burlington, Ontario
  - Milestone Research Inc., London, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Mirtorabi Medicine Professional Corporation, Stouffville, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Manna Research (Toronto), Toronto, Ontario
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- France (2):
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital de La Timone, Marseille
- Germany (12):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - Vitos Orthopaedische Klinik Kassel, Kassel, Hesse
  - Siteworks - Zentrum fur klinische Studien Hannover, Hanover, Lower Saxony
  - Arztepartnerschaft Dr. med. J. Springub/ W. Schwarz -Studienzentrum Nord-West, Westerstede, Lower Saxony
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Universitatsklinikum Jena, Jena, Thuringia
  - Studienzentrum Dr. A Schwittay, Böhlen
  - Datamed GmbH, Cologne
  - Kopfschmerzzentrum Frankfurt, Frankfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Neurologisch-verhaltensmedizinische Schmerzklinik Kiel, Kiel
- Italy (8):
  - Ospedale Sant Andrea - Facolta Medicina Psicologia - Universita degli Studi di Roma Sapienza, Rome, Lazio
  - Fondazione Mondino - Istituto Neurologico Nazionale IRCCS, Pavia, Padua
  - Azienda Ospedaliero Universitaria di Careggi - Cliniche Mediche, Florence, Tuscany
  - IRCCS Istituto delle Scienze Neurologiche Bologna, Unità Operativa di Neurologia - Ospedale Bellaria, Bologna
  - ASST Spedali Civili di Brescia, U.O. Neurologia, Brescia
  - Neurorehabilitation Unit-ICOT Istituto Marco Pasquali, Latina
  - Istituto Neurologico "Carlo Besta" Fondazione IRCCS, Milan
  - IRCCS San Raffaele Roma, Rome
- Poland (14):
  - Solumed Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Krakowska Akademia Neurologii Sp. Z o.o., Krakow, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - Indywidualna Praktyka Lekarska Dr Hab. Med. Anna Szczepanska-Szerej, Lublin, Lublin Voivodeship
  - Next Stage Sp. Z o.o., Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Czestochowa, Częstochowa, Silesian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice, Silesian Voivodeship
  - Neurologia Slaska Centrum Medyczne, Katowice, Silesian Voivodeship
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Spain (7):
  - Neurology Service: Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinico Universitario de Valladolid • HCUV, Valladolid, Castille and León
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Universitario La Paz, Madrid
  - Virgen del Rocio Hospital, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (6):
  - Pharmasite, Malmo, Skåne County
  - CTC Clinical Trial Consultants AB, Stockholm, Stockholms LÄN [se-01]
  - Ladulaas Clinical Trials, Borås
  - ProbarE i Lund, Lund
  - ProbarE i Stockholm AB, Stockholm
  - Studieenheten Akademiskt Specialistcentrum SLSO, Stockholm
- United Kingdom (14):
  - Royal Primary Care Ashgate, Chesterfield Royal Hospital, NHS Foundation Trust, Chesterfield, Derbyshire
  - Panthera Biopartners, Rochdale, Great Manchester
  - Re:Cognition Health - Winchester, Winchester, Hampshire
  - Panthera Bio Partners, Preston, Lancashire
  - Re:Cognition Health - London, London, Marylebone
  - Re:Cognition Health-Private Practice, London, Marylebone
  - Lakeside Healthcare Research, Corby, Northamptonshire
  - CPS Research, Glasgow, Scotland
  - Re-Cognition Health - Bristol, Bristol, South WEST
  - Panthera Biopartners - Sheffield, Sheffield, South Yorkshire
  - Re-Cognition Health, Guildford, Surrey
  - Re-Cognition Health, Birmingham, WEST Midlands
  - Panthera Biopartners Glasgow, Glasgow
  - Panthera Biopartners - Enfield, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1415 participants were enrolled in the study, of which 716 failed screening and 699 participants were randomized. Of the 699 randomized participants, 692 participants received the study intervention.
Groups:
- Double Blind (DB) Rimegepant/ Placebo/ Open Label (OL) Rimegepant: Participants received rimegepant (RMG) 75 mg, orally disintegrating tablets (ODT), once every other day (EOD) alternating with matching placebo dosed EOD for 12 weeks in the double blind treatment (DBT) phase. Eligible participants received RMG 75 mg ODT once daily (QD) for 12 weeks in the open label extension (OLE) phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB Rimegepant/OL Rimegepant: Participants received RMG 75 mg ODT, once daily for 12 weeks in the DBT phase. Eligible participants continued to receive RMG 75 mg ODT once daily for 12 weeks in the OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB Placebo/OL Rimegepant: Participants received matching placebo for RMG 75 mg ODT once daily for 12 weeks, in the DBT phase. Eligible participants received RMG 75 mg ODT once daily for 12 weeks in the OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
Period: DBT Phase
Arm/Group | Double Blind (DB) Rimegepant/ Placebo/ Open Label (OL) Rimegepant | DB Rimegepant/OL Rimegepant | DB Placebo/OL Rimegepant
Started | 234 | 232 | 233
Treated | 232 | 229 | 231
Completed | 204 | 209 | 208
Not Completed | 30 | 23 | 25
Not completed — Adverse Event | 7 | 2 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Protocol-specified withdrawal criterion met | 4 | 6 | 5
Not completed — Withdrawal of consent | 8 | 5 | 7
Not completed — Other | 7 | 3 | 4
Not completed — Randomized, not treated | 2 | 3 | 2
Period: OLE Phase
Arm/Group | Double Blind (DB) Rimegepant/ Placebo/ Open Label (OL) Rimegepant | DB Rimegepant/OL Rimegepant | DB Placebo/OL Rimegepant
Started | 182 (Eligible participants who entered OLE phase.) | 196 (Eligible participants who entered OLE phase.) | 195 (Eligible participants who entered OLE phase.)
Completed | 170 | 187 | 183
Not Completed | 12 | 9 | 12
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Extension phase eligibility failure | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Other | 3 | 5 | 4
Not completed — Withdrawal of consent | 3 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Double-blind treatment safety population included participants in the enrolled analysis set who took greater than equal to (>=) 1 dose of double-blind study drug (rimegepant or placebo).
Groups:
- DB Rimegepant/ Placebo/ OL Rimegepant: Participants received RMG 75 mg ODT, EOD alternating with matching placebo dosed EOD for 12 weeks in the DBT phase. Eligible participants received RMG 75 mg ODT QD for 12 weeks in OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | DB Rimegepant/ Placebo/ OL Rimegepant | DB Rimegepant/OL Rimegepant | DB Placebo/OL Rimegepant | Total
Number analyzed (Participants) | 232 | 229 | 231 | 692
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (11.96) | 43.9 (12.05) | 42.9 (12.35) | 43 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 192 | 207 | 600
  Male | 31 | 37 | 24 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here "Number Analyzed" signifies number of participants evaluable for this baseline characteristic.
  Participants
    number analyzed (Participants) | 70 | 70 | 76 | 216
    Hispanic or Latino | 23 | 20 | 25 | 68
    Not Hispanic or Latino | 47 | 50 | 51 | 148
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here "Number Analyzed" signifies number of participants evaluable for this baseline characteristic.
  Participants
    number analyzed (Participants) | 70 | 70 | 76 | 216
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 5 | 1 | 6 | 12
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
    Black or African American | 6 | 12 | 6 | 24
    White | 56 | 56 | 63 | 175
    More than one race | 0 | 1 | 0 | 1
    Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Observation Phase (OP) in the Number of Migraine Days Per Month Over Entire DBT Phase (Weeks 1 to 12)
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for >=30 minutes, and meeting either >=2 of the pain features: unilateral location; pulsating quality; moderate or severe pain intensity; aggravation by or causing avoidance of routine physical activity OR >=1 of the associated symptoms: nausea and/or vomiting; photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived for a month in on-DBT efficacy analysis period as follows: 28*(total number of migraine days through Month 3 [Weeks 1 to 12]/ (total number of e-diary efficacy data days through Month 3 [Weeks 1 to 12]). Mean change in number of migraine days per month in DBT phase as compared to OP phase was calculated and reported in this outcome measure.
Time Frame: Observation phase (from 31 days prior to randomization), DBT phase (through Month 3 [Week 1 to 12])
Population: Double-blind treatment efficacy (Migraine) analysis set included participants in the full analysis set who were randomized only once and took >= 1 dose of double-blind study drug (rimegepant or placebo) and had >=14 days of eDiary efficacy data (not necessarily consecutive) in both the OP and >=1 month (4-week interval) in the DBT Phase.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Days per month
Groups:
- DB Rimegepant/ Placebo: Participants received RMG 75 mg, ODT, once EOD alternating with matching placebo dosed EOD for 12 weeks in the DBT phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB Rimegepant: Participants received RMG 75 mg ODT, once daily for 12 weeks in the DBT phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB Placebo: Participants received matching placebo for RMG 75 mg ODT once daily for 12 weeks, in the DBT phase. Participants were followed up for 8 weeks after last dose of study drug.
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 221 | 220 | 224
Days per month | -2.9 [-3.31 to -2.42] | -4.0 [-4.44 to -3.60] | -2.2 [-2.65 to -1.85]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; Linear mixed effects model with repeated measures with the number of total migraine days per month in the OP as a covariate; treatment group, randomization stratum (use of previous prophylactic migraine medication generally considered to have efficacy), month and month-by-treatment group interaction as fixed effects; Test type: Superiority; p = 0.0220, Mixed Models Analysis; Least square mean (LSM) Difference = -0.6, 97.5% CI 2-sided [-1.22 to -0.01]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM Difference = -1.8, 97.5% CI 2-sided [-2.35 to -1.19]

2. Secondary Outcome: Percentage of Participants With Greater Than Equal to (>=) 50 Percent (%) Reduction From OP in Number of Moderate to Severe Migraine Days Per Month Over the Entire DBT Phase (Weeks 1 to 12)
Description: Percentage of participants with >= 50% reduction from OP, in number of migraine days (moderate or severe) in the overall DBT phase is reported in this outcome measure. The number of migraine days per month were prorated to 28 days and derived for a month in on-DBT efficacy analysis period as follows: 28*(total number of migraine days through Month 3 [Weeks 1 to 12]/ (total number of e-diary efficacy data days through Month 3 [Weeks 1 to 12]).
Time Frame: DBT phase (through Month 3 [Week 1 to 12])
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 221 | 220 | 224
Percentage of participants | 40.5 [33.5 to 47.9] | 58.1 [50.7 to 65.3] | 33.3 [26.4 to 40.2]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; Mantel-Haenszel risk estimation was used; Test type: Superiority; p = 0.0966, Mantel Haenszel; Difference in percentage = 7.4, 97.5% CI 2-sided [-2.6 to 17.4]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; Mantel-Haenszel risk estimation was used; Test type: Superiority; p < 0.0001, Mantel Haenszel; Difference in percentage = 24.7, 97.5% CI 2-sided [14.6 to 34.8]

3. Secondary Outcome: Mean Change From OP in the Number of Migraine Days Per Month in the Last 4 Weeks (Weeks 9 to 12) of DBT Phase
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for >=30 minutes, and meeting either >=2 of the pain features: unilateral location; pulsating quality; moderate or severe pain intensity; aggravation by or causing avoidance of routine physical activity OR >=1 of the associated symptoms: nausea and/or vomiting; photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived a month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in the month) / (total number of e-diary efficacy data in the month). Mean change in number of migraine days per month in the last 4 weeks of DBT phase as compared to OP phase was calculated and reported in this outcome measure.
Time Frame: Observation phase (from 31 days before randomization), Week 9 to Week 12 of the DBT phase
Population: Double-blind treatment efficacy (Migraine) analysis set included participants in the full analysis set who were randomized only once and took >= 1 dose of double-blind study drug (rimegepant or placebo) and had >=14 days of eDiary efficacy data (not necessarily consecutive) in both the OP and >=1 month (4-week interval) in the DBT Phase. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Days per month
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 203 | 206 | 209
Days per month | -3.0 [-3.59 to -2.49] | -4.2 [-4.75 to -3.75] | -2.8 [-3.33 to -2.33]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; Linear mixed effects model with repeated measures with the number of total migraine days per month in the OP as a covariate; treatment group, randomization stratum (use of previous prophylactic migraine medication generally considered to have efficacy) month and month-by-treatment group interaction as fixed effects; Test type: Superiority; p = 0.5314, Mixed Models Analysis; LS Mean Difference = -0.2, 97.5% CI 2-sided [-0.95 to 0.54]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.4, 97.5% CI 2-sided [-2.12 to -0.71]

4. Secondary Outcome: Mean Change From OP in the Number of Migraine Days Per Month in the First 4 Weeks (Weeks 1 to 4) of DBT Phase
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for >=30 minutes, and meeting either >=2 of the pain features: unilateral location; pulsating quality; moderate or severe pain intensity; aggravation by or causing avoidance of routine physical activity OR >=1 of the associated symptoms: nausea and/or vomiting; photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived a month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in the month / (total number of e-diary efficacy data in the month. Mean change in number of migraine days per month in the first 4 weeks of DBT phase as compared to OP phase was calculated and reported in this outcome measure.
Time Frame: Observation phase (from 31 days before randomization), Week 1 to Week 4 of the DBT phase
Population: as for outcome 3
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Days per month
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 220 | 219 | 224
Days per month | -2.7 [-3.17 to -2.16] | -3.6 [-4.10 to -3.16] | -1.5 [-1.97 to -1.05]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS Mean Difference = -1.2, 97.5% CI 2-sided [-1.84 to -0.47]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.1, 97.5% CI 2-sided [-2.78 to -1.46]

5. Secondary Outcome: Mean Number of Acute Migraine-Specific Medication Days Per Month Over the Entire DBT Phase (Weeks 1 to 12)
Description: An acute migraine-specific medication day was defined as any calendar day during which the participant took a migraine-specific medication (i.e., triptan or ergotamine). The number of acute migraine-specific medication days per month were prorated to 28 days and derived for on-DBT efficacy analysis period as follows: 28*(total number of acute migraine-specific medication days through Month 3/ (total number of e-Diary efficacy data days through Month 3).
Time Frame: DBT phase (through Month 3 [Week 1 to 12])
Population: as for outcome 1
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Days per month
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 221 | 220 | 224
Days per month | 2.3 [1.87 to 2.82] | 1.5 [1.13 to 1.88] | 2.8 [2.28 to 3.35]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; Linear mixed effects model with repeated measures has treatment group, randomization stratum, month, and month-by-treatment group interaction as fixed effects; Test type: Superiority; p = 0.1440, Mixed Models Analysis; LS Mean Difference = -0.5, 97.5% CI 2-sided [-1.20 to 0.25]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.3, 97.5% CI 2-sided [-1.97 to -0.65]

6. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality-of-Life Questionnaire (MSQoL) Version 2.1 Restrictive Role Function Domain Score at Week 12 of the DBT Phase
Description: MSQoL is a self-administered, 14-item instrument validated in 3 domains: role restriction, role prevention, and the emotional function. The restrictive role function domain consisted of 7 items that described how migraine limited one's daily social and work-related activities. Participants were required to respond to items using a 6-point scale ranging from 1 to 6, where "1: none of the time," "2: a little bit of the time," "3: some of the time," "4: a good bit of the time," "5: most of the time," and "6: all of the time,". Item scores were recoded using (7 - original score). Raw dimension scores for restrictive role function domain were computed as a sum of recoded item scores and rescaled from a 0 to 100 scale such that lower score (0) indicated poor quality of life and higher scores (100) indicated better quality of life.
Time Frame: Baseline (Day 1), Week 12 of the DBT phase
Population: Double-blind treatment efficacy analysis set included participants in the full analysis set who were randomized only once and took >= 1 dose of double-blind study drug. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Units on a scale
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 194 | 191 | 197
Units on a scale | 21.3 [18.37 to 24.33] | 29.1 [25.79 to 32.31] | 18.9 [15.91 to 21.97]
Statistical Analysis 1: Comparison: DB Rimegepant/ Placebo vs DB Placebo; Linear regression model with treatment group and randomization stratum as fixed effects and baseline score as covariate for participants with non-missing domain scores at both baseline and Week 12; Test type: Superiority; p = 0.2029, Regression, Linear; LS Mean Difference = 2.4, 97.5% CI 2-sided [-1.84 to 6.66]
Statistical Analysis 2: Comparison: DB Rimegepant vs DB Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Linear; LS Mean Difference = 10.1, 97.5% CI 2-sided [5.71 to 14.52]

7. Secondary Outcome: Number of Participants With Mild, Moderate and Severe Adverse Events (AEs) in DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. AEs were categorized as mild: usually transient and required only minimal treatment or therapeutic intervention. The event did not generally interfere with usual activities of daily living. Moderate: was usually alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but posed no significant or permanent risk of harm to the participant. Severe: Interrupted usual activities of daily living, significantly affected clinical status, or required intensive therapeutic intervention. AEs included both non-SAEs and serious adverse events (SAEs).
Time Frame: DBT: From Week 1 to Week 20
Population: Double-blind treatment safety population included participants in the enrolled analysis set who took >= 1 dose of double-blind study drug (rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants
  Mild | 73 | 86 | 91
  Moderate | 42 | 22 | 43
  Severe | 4 | 3 | 2

8. Secondary Outcome: Number of Participants With Mild, Moderate and Severe AEs OLE Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. AEs were categorized as mild: usually transient and required only minimal treatment or therapeutic intervention. The event did not generally interfere with usual activities of daily living. Moderate: was usually alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but posed no significant or permanent risk of harm to the participant. Severe: Interrupted usual activities of daily living, significantly affected clinical status, or required intensive therapeutic intervention. AEs included both non-SAEs and SAEs.
Time Frame: OLE: From Week 12 to Week 32
Population: Open-label rimegepant safety population included participants in the enrolled analysis set who took >= 1 dose of open-label rimegepant.
Measure: Count of Participants; unit: Participants
Groups:
- DB RMG EOD/DB PBO EOD/ OL RMG QD: Participants who received RMG 75 mg, ODT alternating with matching placebo in the DBT phase received RMG 75 mg ODT QD for 12 weeks in the OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB RMG QD/ OL RMG QD: Participants who received RMG 75 mg ODT in the DBT phase continued to receive RMG 75 mg ODT once daily for 12 weeks in the OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
- DB PBO QD/ OL RMG QD: Participants who received placebo ODT in the DBT phase received RMG 75 mg ODT once daily for 12 weeks in the OLE phase. Participants were followed up for 8 weeks after last dose of study drug.
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants
  Mild | 65 | 57 | 65
  Moderate | 30 | 22 | 25
  Severe | 2 | 2 | 1

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. An SAE was any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of the participant who received rimegepant and other important medical events.
Time Frame: DBT: From Week 1 to Week 20
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants | 3 | 2 | 1

10. Secondary Outcome: Number of Participants With SAEs in OLE Phase
Description: as for outcome 9
Time Frame: OLE: From Week 12 to Week 32
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants | 2 | 2 | 2

11. Secondary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation in DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. In this outcome measure, participants with adverse events leading to study drug discontinuation were reported.
Time Frame: DBT: From Week 1 to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants | 6 | 1 | 4

12. Secondary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation in OLE Phase
Description: as for outcome 11
Time Frame: OLE: From Week 12 to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants | 4 | 1 | 1

13. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in DBT Phase
Description: The laboratory parameters were graded according to the National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 and using division of AIDS (DAIDS) toxicity grading scale version 2.1 (glucose, low density lipoprotein [LDL] cholesterol, uric acid and urinalysis) and for other parameters (eosinophils, hemoglobin, leukocytes, albumin, lymphocytes, neutrophils, platelets, alanine aminotransferase, alkaline phosphatase ,aspartate aminotransferase, bicarbonate, bilirubin, calcium, cholesterol, creatine kinase, creatinine, lactate dehydrogenase, potassium, sodium, triglycerides) CTCAE version v5.0 was used. Severity were graded as Grade 1=mild AE, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening consequences; urgent intervention indicated. Number of participants according to Grade 3 or 4 laboratory abnormalities are reported. Only laboratory abnormalities with non-zero values in any of the treatment arms are reported.
Time Frame: DBT: From Week 1 to Week 20
Population: Double-blind treatment safety population included participants in the enrolled analysis set who took >= 1 dose of double-blind study drug (rimegepant or placebo). All participants under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants
  Lymphocytes, low: number analyzed (Participants) | 225 | 224 | 224
  Lymphocytes, low | 0 | 0 | 1
  Alanine Aminotransferase: number analyzed (Participants) | 225 | 224 | 225
  Alanine Aminotransferase | 0 | 1 | 1
  Aspartate Aminotransferase: number analyzed (Participants) | 225 | 224 | 225
  Aspartate Aminotransferase | 0 | 0 | 1
  Creatine Kinase: number analyzed (Participants) | 225 | 224 | 225
  Creatine Kinase | 2 | 1 | 4
  Glucose, low: number analyzed (Participants) | 225 | 224 | 225
  Glucose, low | 0 | 1 | 0
  LDL Cholesterol: number analyzed (Participants) | 207 | 213 | 218
  LDL Cholesterol | 6 | 4 | 9
  LDL Cholesterol, fasting: number analyzed (Participants) | 107 | 120 | 118
  LDL Cholesterol, fasting | 4 | 3 | 3
  LDL Cholesterol, not fasting: number analyzed (Participants) | 102 | 96 | 102
  LDL Cholesterol, not fasting | 2 | 1 | 6
  Sodium, high: number analyzed (Participants) | 225 | 224 | 225
  Sodium, high | 0 | 0 | 1
  Triglycerides: number analyzed (Participants) | 207 | 213 | 218
  Triglycerides | 0 | 1 | 0
  Triglycerides, fasting: number analyzed (Participants) | 107 | 120 | 118
  Triglycerides, fasting | 0 | 1 | 0
  Urinalysis Glucose: number analyzed (Participants) | 204 | 207 | 213
  Urinalysis Glucose | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in OLE Phase
Description: The laboratory parameters were graded according to the NCI CTCAE version 5.0 and using DAIDS toxicity grading scale version 2.1 (glucose, LDL cholesterol, uric acid and urinalysis). And for other parameters (eosinophils, hemoglobin, leukocytes, albumin, lymphocytes, neutrophils, platelets, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, calcium, cholesterol, creatine kinase, creatinine, lactate dehydrogenase, potassium, sodium, triglycerides) CTCAE version v5.0 was used. Severity was graded as Grade 1=mild AE, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening consequences; urgent intervention indicated. Number of participants according to Grade 3 or 4 laboratory abnormalities are reported. Only laboratory abnormalities with non-zero values in any of the treatment arms are reported.
Time Frame: OLE: From Week 12 to Week 32
Population: Open-label rimegepant safety population included participants in the enrolled analysis set who took >= 1 dose of open-label rimegepant. All participants under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants
  Alanine Aminotransferase: number analyzed (Participants) | 180 | 193 | 194
  Alanine Aminotransferase | 1 | 1 | 1
  Aspartate Aminotransferase: number analyzed (Participants) | 180 | 193 | 194
  Aspartate Aminotransferase | 0 | 1 | 0
  Creatine Kinase: number analyzed (Participants) | 180 | 191 | 190
  Creatine Kinase | 3 | 0 | 5
  LDL Cholesterol: number analyzed (Participants) | 166 | 182 | 179
  LDL Cholesterol | 7 | 8 | 4
  LDL Cholesterol, fasting: number analyzed (Participants) | 80 | 101 | 88
  LDL Cholesterol, fasting | 4 | 4 | 0
  LDL Cholesterol, not fasting: number analyzed (Participants) | 89 | 81 | 92
  LDL Cholesterol, not fasting | 3 | 4 | 4
  Potassium, low: number analyzed (Participants) | 180 | 191 | 190
  Potassium, low | 0 | 1 | 0
  Potassium, high: number analyzed (Participants) | 180 | 191 | 190
  Potassium, high | 1 | 0 | 1
  Triglycerides: number analyzed (Participants) | 166 | 182 | 179
  Triglycerides | 0 | 1 | 0
  Triglycerides, not fasting: number analyzed (Participants) | 89 | 81 | 92
  Triglycerides, not fasting | 0 | 1 | 0
  Urinalysis Glucose: number analyzed (Participants) | 162 | 176 | 175
  Urinalysis Glucose | 1 | 1 | 0

15. Secondary Outcome: Number of Participants With Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) Elevations > 3* Upper Limit of Normal (ULN) Concurrent With (Total Bilirubin) TBL >2*ULN in DBT Phase
Description: Number of participants with AST or ALT >3*ULN concurrent with TBL >2*ULN in DBT phase were reported in this outcome measure.
Time Frame: DBT: From Week 1 to Week 20
Population: Double-blind treatment safety population included participants in the enrolled analysis set who took >= 1 dose of double-blind study drug (rimegepant or placebo). Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 225 | 224 | 225
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With AST or ALT Elevations > 3* ULN Concurrent With TBL >2*ULN in OLE Phase
Description: as for outcome 15
Time Frame: OLE: From Week 12 to Week 32
Population: Open-label rimegepant safety population included participants in the enrolled analysis set who took >= 1 dose of open-label rimegepant. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 180 | 193 | 194
Participants | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Hepatic-Related AEs in the DBT Phase
Description: \An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. Hepatic-related AEs included: alanine aminotransferase and aspartate aminotransferase increased, liver function test abnormal, liver function test increased, bilirubin conjugated increased, blood bilirubin increased, transaminases increased and hyperbilirubinemia. Number of participants with any hepatic-related AEs in the DBT phase were reported in this outcome measure.
Time Frame: DBT: From Week 1 to Week 20
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants | 7 | 8 | 8

18. Secondary Outcome: Number of Participants With Hepatic-Related AEs in the OLE Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. Hepatic AEs included: alanine aminotransferase and aspartate aminotransferase increased, liver function test abnormal, bilirubin conjugated, hepatic enzyme increased, blood bilirubin unconjugated increased, blood bilirubin and transaminases increased and hepatic function abnormal. Number of participants with any hepatic-related AEs in the OLE phase were reported in this outcome measure.
Time Frame: OLE: From Week 12 to Week 32
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants | 11 | 4 | 6

19. Secondary Outcome: Number of Participants With Hepatic-Related AEs Leading to Study Drug Discontinuation in the DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. Hepatic-related AEs included: alanine aminotransferase and aspartate aminotransferase increased, liver function test and blood bilirubin increased. Number of participants with any hepatic-related AEs leading to study drug discontinuation is reported in this outcome measure.
Time Frame: DBT: From Week 1 to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo
Number analyzed (Participants) | 232 | 229 | 231
Participants | 4 | 1 | 2

20. Secondary Outcome: Number of Participants With Hepatic-Related AEs Leading to Study Drug Discontinuation in the OLE Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. Hepatic-related AEs included: aspartate aminotransferase increased and liver function test abnormal. Number of participants with any hepatic-related AEs leading to study drug discontinuation is reported in this outcome measure.
Time Frame: OLE: From Week 12 to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
Number analyzed (Participants) | 182 | 196 | 195
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks after last dose of study drug (DBT phase: Week 1 to Week 20; OLE phase Week 12 to Week 32)
Description: Same event may appear as AE and SAE, but what is presented are distinct events. Event may be categorized as serious in 1 and as non-SAE in another participant, or 1 participant may have experienced both serious and non-SAE.DB treatment safety population=participants in the enrolled analysis set who took>=1 dose of DB study drug (rimegepant or placebo) used for DBT phase arms. OL RMG safety population included participants in the enrolled analysis set who took >= 1 dose of open-label rimegepant.
Arm/Group | DB Rimegepant/ Placebo | DB Rimegepant | DB Placebo | DB RMG EOD/DB PBO EOD/ OL RMG QD | DB RMG QD/ OL RMG QD | DB PBO QD/ OL RMG QD
All-Cause Mortality (participants affected / at risk) | 0/232 | 0/229 | 0/231 | 0/182 | 0/196 | 0/195
Serious Adverse Events (participants affected / at risk) | 3/232 | 2/229 | 1/231 | 2/182 | 2/196 | 2/195
Other Adverse Events (participants affected / at risk) | 13/232 | 13/229 | 13/231 | 17/182 | 19/196 | 13/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Rimegepant/ Placebo (N=232) | DB Rimegepant (N=229) | DB Placebo (N=231) | DB RMG EOD/DB PBO EOD/ OL RMG QD (N=182) | DB RMG QD/ OL RMG QD (N=196) | DB PBO QD/ OL RMG QD (N=195)
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Status migrainosus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Rimegepant/ Placebo (N=232) | DB Rimegepant (N=229) | DB Placebo (N=231) | DB RMG EOD/DB PBO EOD/ OL RMG QD (N=182) | DB RMG QD/ OL RMG QD (N=196) | DB PBO QD/ OL RMG QD (N=195)
Nasopharyngitis (Infections and infestations) | 13 | 13 | 13 | 13 | 5 | 7
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 4 | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT05217927/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05217927/SAP_001.pdf